CLINICAL TRIAL: NCT02720874
Title: Multidisciplinary Approach to Patient-Physician Partnership In Treating To Target In Rheumatoid Arthritis
Brief Title: Multidisciplinary Approach for Treat To Target In Rheumatoid Arthritis
Acronym: MAPPIT-RA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, George A Karpouzas, MD, Associate Professor of Medicine, UCLA, Chief, Division of Rheumatolgy, Harbor-UCLA Medical Center, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21625-01
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): In the multifaceted intervention, participants will first receive an educational session with monthly follow-up phone calls from a trained rheumatology nurse. A rheumatoid arthritis educational booklet will also be provided. During regularly scheduled clinic appointments (at baseline, 3 months, 6 months, 9 months, and 12 months), participants will receive multidisciplinary rheumatologic care, including evaluation by a rheumatologist, physical therapist and psychologist. In addition, participants will be scheduled for ad hoc rheumatology appointments if technology-based symptom monitoring and reporting indicates a marked increase in RA disease activity.
  Interventions: Behavioral: Rheumatoid arthritis educational booklet; Behavioral: Multidisciplinary rheumatologic care; Behavioral: Nurse education and monthly calls; Behavioral: Technology-based symptom monitoring and reporting
- Control Arm (Active Comparator): Participants will receive standard of care treatment from their assigned rheumatologists during routine clinic appointments scheduled quarterly for the 12-month trial duration. Referrals to ancillary services will occur in a standard of care fashion. Participants will additionally receive monthly healthcare coordinator calls and be given the rheumatoid arthritis educational booklet.
  Interventions: Behavioral: Rheumatoid arthritis educational booklet; Behavioral: Monthly healthcare coordinator calls

INTERVENTIONS:
Behavioral: Rheumatoid arthritis educational booklet — Participants will receive a low-literacy rheumatoid arthritis educational booklet that provides general disease state information.
Behavioral: Multidisciplinary rheumatologic care — At each regularly scheduled clinic appointment, participants will receive treatment from their assigned rheumatologist, undergo an in-clinic physical therapy evaluation and, if indicated, a psychological evaluation. Physical therapy and psychology follow-up sessions will occur as directed by the individual services.
  Arms: Intervention Arm
Behavioral: Nurse education and monthly calls — Participants will meet one-on-one with a rheumatology nurse for a tailored educational session encompassing disease state education, an introduction of the treat to target concept, an overview of treatment options, and goal setting and planning. During monthly follow-up calls, participant educational needs will be addressed; goal setting, planning and review will also be conducted.
  Arms: Intervention Arm
Behavioral: Monthly healthcare coordinator calls — During monthly calls with the healthcare coordinator, specific questions and concerns raised by participants may be addressed. The primary purpose of these calls is to control for potential benefit derived from time on the phone with a health professional.
  Arms: Control Arm
Behavioral: Technology-based symptom monitoring and reporting — When at home patient self-monitoring reports indicate a significant increase in RA disease activity, participants will be promptly contacted and scheduled for an ad hoc evaluation with their treating rheumatologist.
  Arms: Intervention Arm

SUMMARY:
This research will evaluate a multifaceted patient-centered intervention in a sample of socioeconomically disadvantaged Hispanic adults with rheumatoid arthritis (RA) that capitalizes on a partnership between the extended rheumatology healthcare team and each patient in order to promote understanding, uptake and adherence to the principles of treat-to-target strategy. The primary hypothesis of this study is that the addition of a multifaceted intervention incorporating integrated multidisciplinary rheumatologic care, nurse-directed self-management education and supportive follow-up, and technology-based at home RA symptom monitoring and reporting to clinical guideline-based care will increase RA remission rate at 6 months.

DETAILED DESCRIPTION:
One hundred and fifty Hispanic RA patients will be recruited for this proposal and randomized 1:1 to Intervention and Control arms for a period of 12 months. Participants will be recruited from the Adult Rheumatology clinic at Harbor-UCLA. Patients who meet enrollment criteria based on review of electronic medical records will be provided information about the study during regular outpatient visits. Interested patients will be formally screened.

After providing informed consent, eligible patients will complete baseline measures and be randomly assigned into Intervention and Control arms using a minimization protocol, with a goal of enrolling 150 patients (75 in each group). All participants will attend rheumatology clinic appointments scheduled quarterly for the 12-month trial duration, during which they will also complete assessments (at 3, 6, 9, and 12 months post-baseline; see description of outcomes for full detail). Between appointments with their assigned rheumatologist, participants will regularly self-monitor their RA symptoms using the Routine Assessment Patient Index Data (RAPID3) questionnaire administered via an interactive voice response (IVR) phone survey weekly for 12 months.

At baseline, participants will be enrolled in the IVR system and the study coordinator will provide a detailed orientation to the automated phone survey as well as written instructions including the toll-free phone number, and a unique study personal identification number. Participants will each select the day and the hours between which they will complete the weekly phone survey. After entering their unique study personal identification number, participants will complete the 12-item RAPID3 questionnaire, entering responses using their telephone keypad. If they do not call in and complete the survey on their preselected day during the specified time frame, they will receive a reminder call an hour later from the time by which they would have been expected to call in.

At the baseline visit, all participants will receive a rheumatoid arthritis educational booklet that provides general disease state information, including an overview of RA (e.g., its causes, associated symptoms, how it is diagnosed), RA medications and other treatment options, pain management, physical activity, nutrition and diet. The material is written at a sixth grade reading level and incorporates simple figures and graphics to enhance readability and promote participant comprehension and engagement. The study coordinator will also give each participant a pedometer and provide instruction for its use. Participants will be encouraged to wear the pedometer during waking hours and record their total daily steps in a log, along with the type and duration of other activities like swimming that pedometers do not capture.

Control arm participants will receive standard of care treatment from their assigned rheumatologists. Pharmacotherapy will be monitored and adjusted by the treating rheumatologist in accordance with evidence-based clinical practice guidelines. Physical Therapy referrals and evaluations will occur as indicated for addressing specific problems. Referral for psychological services will be provided when patients endorse symptoms of depression in response to a verbal screen or participant-initiated discussion. Control arm participants will also have regularly scheduled 20-30 minute monthly phone calls with the healthcare coordinator. While questions and concerns specifically raised by participants regarding study procedure and the content of the educational booklet will be addressed, these phone calls are primarily designed to control for potential benefit participants may derive from time on the phone with a health professional. The healthcare coordinator will engage participants using a non-directive approach based on use of active listening, reflective statements and similar techniques.

Intervention arm participants will receive integrated treatment from a multidisciplinary healthcare team during the routine clinic visits. In addition to appointments with their assigned rheumatologist, a physical therapist will assess participants' physical functioning, provide joint protection guidance and assist patients in making physical fitness plans based on their own goals and tailored to patients' abilities and physical limitations. Interim individual physical therapy sessions will be scheduled in accordance with the physical therapist's recommendations. Additionally, if during any routine clinic appointment a participant scores 10 or higher on the PHQ-9 and/or endorses symptoms of depression in response to a verbal screen, they will receive a same-day, in-clinic psychological evaluation. The psychologist will assess whether patient symptoms meet diagnostic criteria for a depressive disorder and, when clinically indicated, provide recommendations for treatment. Follow-up treatment appointments will be scheduled with patients by the psychologist.

In addition to regularly scheduled rheumatology appointments, if between-visit patient self-monitoring reports indicate an increase in RA disease activity (flare), participants in the intervention arm will be scheduled for an ad hoc evaluation with their assigned rheumatologist. Specifically, if participants' RAPID3 surveys show two consecutive week-to-week score increases and the cumulative two week RAPID3 increase is greater than 1.2 points, they will be contacted by the study coordinator that day (or following morning if surveys are completed after regular office hours) to schedule an ad-hoc appointment with their rheumatologist within 2 working days. During routine and ad hoc intervention arm patient visits, while clinical practice guidelines will inform rheumatologist monitoring of pharmacotherapy, the treatment planning process will be grounded in a shared decision making framework.

Participants in the intervention arm will further be provided a one-on-one tailored education session with a trained rheumatology nurse that will encompass a general disease state education, incorporating pictograms and short slide presentations, an introduction of the treat to target concept, overview of treatment options, and discussion of patient priorities and identification of personally salient long-term treatment-related goals. During regularly scheduled 20-30 minute monthly follow-up phone calls with each intervention arm participant, the rheumatology nurse will address individual educational needs, answer questions and reinforce learning. Goal setting, planning and review will also be conducted. Specifically, participants will select goals to be achieved in the upcoming month and be assisted in developing specific action plans. The rheumatology nurse will also check in about their work and progress on action plans discussed in the last phone call. Any barriers encountered will be explored and participants will be engaged in a problem-solving process, revising existing action plans as needed.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Greater Los Angeles area and receive rheumatologic care at the adult rheumatology clinic at Harbor-UCLA Medical Center in Torrance, California
* Fulfill the 2010 American College of Rheumatology revised diagnostic criteria for RA
* Have at least moderate disease activity as indicated by a Clinical Disease Activity Index (CDAI) score >10 and Routine Assessment Patient Index Data (RAPID3) score >2
* Be able and willing to provide written informed consent and to adhere to the study visit schedule and other protocol
* Availability of a touch-tone landline or mobile telephone
* Of self-identified Hispanic/Latino descent

Exclusion Criteria:

* Known irreversible articular damage, including subluxations, arthrodesis, fusion, or prosthesis
* Functional class IV as defined by the American College of Rheumatology Classification of Functional Status in rheumatoid arthritis
* Overlapping autoimmune or mixed connective tissue syndromes
* Serious medical conditions, including: chronic infection, advanced or decompensated heart failure, higher than class II chronic kidney disease, cancer (unless in remission for period of 5 years or more), or any uncontrolled medical condition that is deemed by the investigators to interfere with the study protocol
* At risk for suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving remission based on the Clinical Disease Activity Index at 6 months | 6 months
  Remission as defined by a Clinical Disease Activity Index (CDAI) score ≤ 2.8. The CDAI is a pooled disease activity index based on the swollen joint count (0-28), tender joint count (0-28), patient global estimate (0-10), and physician global estimate (0-10); the CDAI scale ranges from 0-76, where higher scores represent higher disease activity.
Percentage of participants achieving remission based on the Routine Assessment Patient Index Data at 6 months | 6 months
  Remission as defined by a Routine Assessment Patient Index Data (RAPID3) score ≤ 1. The RAPID3 is a self-report measure of disease activity and represents the average of patient ratings for physical function, pain and disease activity. Total RAPID3 scores range from 0 to 10, where higher scores represent higher patient-rated disease activity.

SECONDARY OUTCOMES:
Percentage of participants achieving remission based on the Clinical Disease Activity Index at 12 months | 12 months
  Remission as defined by a Clinical Disease Activity Index (CDAI) score ≤ 2.8.
Percentage of participants achieving remission based on the Routine Assessment Patient Index Data at 12 months | 12 months
  Remission as defined by a Routine Assessment Patient Index Data (RAPID3) score ≤ 1.
Percentage of participants with low disease activity based on the Clinical Disease Activity Index | 6 months, 12 months
  Low disease activity defined by a Clinical Disease Activity Index (CDAI) score of 2.81-10.
Percentage of participants with low disease activity based on the Routine Assessment Patient Index Data | 6 months, 12 months
  Low disease activity defined by a Routine Assessment Patient Index Data (RAPID3) score of 1.01-2.
Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) from baseline | Baseline, 3 months, 6 months, 9 months, 12 months
  The HAQ-DI consists of 20 questions measuring patients' self-reported ability to perform activities of daily living in eight functional domains - dressing, arising, eating, walking, hygiene, reach, grip, and usual activities. Scores in each domain range from 0 (no disability) to 3 (completely disabled) and are averaged to calculate the HAQ-DI total score. Higher scores represent higher levels of disability, and negative change scores (visit minus baseline) indicate improvement.
Change in Patient Health Questionnaire (PHQ-9) depression from baseline | Baseline, 3 months, 6 months, 9 months, 12 months
  The PHQ-9 consists of nine items that parallel the diagnostic criteria for major depression in the fourth and fifth editions of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV and DSM-5). Items measure symptoms that have occurred over the past two weeks and are rated on a 4-point scale ranging from 0 (absence of symptoms) to 3 (presence of symptoms nearly every day). Negative change scores (visit minus baseline) indicate improvement.
Change in Patient Global Assessment of disease activity (PGA) from baseline | Baseline, 3 months, 6 months, 9 months, 12 months
  PGA of disease activity is measured using a 10 cm horizontal line visual analog scale. Higher scores represent higher patient-rated rheumatoid arthritis disease activity, and negative change scores (visit minus baseline) indicate improvement.
Change in Pain Visual Analogue Scale (VAS) from baseline | Baseline, 3 months, 6 months, 9 months, 12 months
  The pain VAS asks patients to rate the severity of their arthritis-related pain using a 10 cm horizontal line VAS ranging from no pain (0 cm) to unbearable pain (10 cm). Negative change scores (visit minus baseline) indicate improvement.
Change in Fatigue Visual Analogue Scale (VAS) from baseline | Baseline, 3 months, 6 months, 9 months, 12 months
  The fatigue VAS asks patients to rate the severity of their fatigue over the past week using a 10 cm horizontal line VAS ranging from no fatigue (0 cm) to extreme fatigue (10 cm). Negative change scores (visit minus baseline) indicate improvement.
Change in SF-36 health status from baseline | Baseline, 3 months, 6 months, 9 months, 12 months
  The 36-Item Short-Form Health Survey (SF-36) assesses general health status across eight domains: physical functioning, role limitations-physical, bodily pain, vitality, social functioning, role limitations-emotional, mental health, and general health. These domains can also be summarized as Physical Component Summary and Mental Component Summary scores. SF-36 domain and component summary scores are recalibrated to a 0-100 scale with higher scores indicating better health status; positive change scores (visit minus baseline) indicate improvement.
Change in Rheumatoid Arthritis Specific Work Productivity Survey (WPS-RA) from baseline | Baseline, 3 months, 6 months, 9 months, 12 months
  The WPS-RA is a nine-item questionnaire that assesses the impact of RA on work and household productivity, and participation in daily activities. Employed participants indicate number of work absences (absenteeism) and days with work productivity reduced ≥ 50% (presenteeism). All participants report number of days with no household work performed, days with household productivity reduced ≥ 50%, days that outside help was hired, and days with missed family, social or leisure activities. Participants also rate the extent to which RA interferes with their paid work (if applicable) and household productivity on a 0-10 scale ranging from no interference to complete interference. For all items, negative change scores (visit minus baseline) indicate improvement.

OTHER OUTCOMES:
Brief Illness Perception Questionnaire (BIPQ) | Baseline, 6 months, 12 months
Single Item Health Literacy Screener (SILS) | Baseline, 6 months, 12 months
Patient Knowledge Questionnaire in Rheumatoid Arthritis (PKQ-RA) | Baseline, 6 months, 12 months
Simplified Medication Adherence Questionnaire (SMAQ) | Baseline, 6 months, 12 months
Health Education Impact Questionnaire (heiQ) | Baseline, 6 months, 12 months
Shared Decision Making Questionnaire (SDM-Q-9) | Baseline, 3 months, 6 months, 9 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: George A Karpouzas, MD, Principal Investigator — The Lundquist Institute at Harbor-UCLA Medical Center
Locations (1):
- The Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No